CLINICAL TRIAL: NCT05208632
Title: Perfusion Index and Pleth Variability Index an Early Indicator of the Success of Brachial Plexus Block; Randomized Clinical Triall
Status: Completed | Type: Observational
Sponsor: Malatya Egitim Ve Arastirma Hastanesi (Other Government)
Responsible Party: Principal Investigator, Erdinç Koca, ANESTHESIOLOGY AND REANIMATION CLINIC, Malatya Egitim Ve Arastirma Hastanesi
Other Study IDs: 123456
Record Dates: First submitted 2021-12-13; First posted 2022-01-26 (Actual); Last update posted 2022-01-26 (Actual); Status verified 2022-01

CONDITIONS: Perfusion Index and Pleth Variability Index an Early Indicator of the Success of Brachial Plexus Block; Randomized Clinical Trial
Keywords: brachial plexus; interscalene block; infraclavicular block; Perfusion index; Pleth Variability Index; regional anesthesia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- BLOCK SİDE: 40 patients, including ASA1-2, 20 patients over the age of 18, who were planned for upper extremity surgery, in the interscalen group, and 20 in the supraclavicular group, were included in the study. Demographic data of the patients were recorded by measuring PI and PVI values at baseline before the block and at the 1st, 5th, 10th, 15th, and 20th minutes after the block, both simultaneously.
  Interventions: Other: INTERSCALEN BLOCK APPLICATION WITH USG
- UNBLOCK SİDE: 40 patients, including ASA1-2, 20 patients over the age of 18, who were planned for upper extremity surgery, in the interscalen group, and 20 in the supraclavicular group, were included in the study. Demographic data of the patients were recorded by measuring PI and PVI values at baseline before the block and at the 1st, 5th, 10th, 15th, and 20th minutes after the block, both simultaneously.
  Interventions: Other: INTERSCALEN BLOCK APPLICATION WITH USG

INTERVENTIONS:
Other: INTERSCALEN BLOCK APPLICATION WITH USG — 40 patients, including ASA1-2, 20 patients over the age of 18, who were planned for upper extremity surgery, in the interscalen group, and 20 in the supraclavicular group, were included in the study. Demographic data of the patients were recorded by measuring PI and PVI values at baseline before the block and at the 1st, 5th, 10th, 15th, and 20th minutes after the block, both simultaneously.
  Other Names: SHOULDER SURGERY

SUMMARY:
Abstract:

Background: In investigators study, we aimed to compare PI and PVI between the interscalen block and infraclavicular block and evaluate its use as an early marker in block success.

Meterial- Methods: 40 patients, including ASA1-2, 20 patients over the age of 18, who were planned for upper extremity surgery, in the interscalen group, and 20 in the supraclavicular group, were included in the study. Demographic data of the patients were recorded by measuring PI and PVI values at baseline before the block and at the 1st, 5th, 10th, 15th, and 20th minutes after the block, both simultaneously.

DETAILED DESCRIPTION:
investigators study, which was designed as a prospective clinical study, was initiated in accordance with the according to the consort flow diagram, after the approval of the clinical research ethics committee of Malatya Turgut Özal University, dated 03.08.2021 and numbered 2021/43. investigators study was carried out in accordance with the Helsinki declaration published in 2013.The patients were randomly divided into two groups as the patients who underwent interscalen block (ISB) and infraclavicular block (ICB) by the closed-envelope method by a blind nurse who did not participate in the study. Based on similar studies, the sample size of the study was calculated as 0.05 patients with alpha and 0.8 patients with a beta, 20 patients in each group, a total of 40 patients. 46 patients over the age of 18 with ASA classification (American Society of Anesthesiologists) I-II, who were planned to undergo upper extremity surgery, were included in the study. 6 patients were excluded from the study because they were switched to general anesthesia, and 40 patients who developed successful block were included in the study. Pediatric patients, pregnant patients, patients with peripheral arterial disease, heart failure with a hemoglobin level of 10, renal failure, liver failure, coagulation disorder with neuropathy, and patients with known allergy to local anesthetics were excluded from the study. Wet signed informed consent was obtained from all patients.

All patients included in the study were examined by an anesthesiologist before anesthesia. Following the appropriate fasting period, the patients were taken to the preparation room and routine monitoring (peripheral oxygen saturation, non-invasive arterial measurement of blood pressure and Electrocardiogram) were performed. Vascular access was established with a 20G branule in the other arm, which did not undergo surgery. The patients were administered midazolam (0.05-0.1 mg/kg, Dormicum 5mg/5cc, Deva İlaç, Istanbul) for sedation before the procedure. Nasal oxygen was given at 2-4 L/min. In addition to routine monitoring, both upper extremities Perfusion index: PI, Plethysmographic variability index: PVI, hemoglobin HGB, (The probe of a MasimoRadical 7, MasimoCorp. Irvine, CA, USA) were performed. Using an insulated neurostimulation needle (22 G, 50 mm Locoplex, Vygon®, France) accompanied by USG (Samsung HM70 Evo, South Korea) and nerve stimulator (Stimuplex, HNS 11; Braun Melsunçgen, Melsungen, Germany) Interscalen block was performed in 20 patients and the infraclavicular block were performed in 20 patients. After turning the head to the opposite side of the patients in the interscalen group, a skin anti setting was provided with povidone-iodine in the treatment area. The USG probe was placed transversely obliquely from the level of the cricoid cartilage (C6) to the line connecting the interscalen space and the brachial plexus was found and 22G 50 mm insulated nerve stimulator needle was inserted in-plain with a posterior approach and 10 mL of 0.5% bupivacaine, 10 mL of 2% lidocaine, 10 mL of 2% prilocaine were injected considering the loss of response at currents less than 0.2-0.3 mA to avoid the risk of intraneural injection after a distal motor response was found at <0.5 mA with a nerve stimulator. In the infraclavicular group, after the area was cleaned with povidone-iodine, the USG probe was placed in the area where the clavicle and the cricoid process intersect, and the anatomical structure was observed. A 22G 50 mm stimulator needle was inserted with the in-plain approach, and after the distal motor response was found at < 0.5 mA with the nerve stimulator, to avoid the risk of intraneural injection, considering the loss of response at currents less than 0.2-0.3 mA, 10 mL % 0.5 bupivacaine, 10 ml 2% lidocaine, 10 ml 2% prilocaine injections were administered. The development of sensorineural block (inability to identify the cold application) in the motor block and related dermatomes was accepted as a successful block.

Demographic data such as age, gender, height, weight, and body mass index (BMI) of the patients and entry hemoglobin levels were recorded. Heart rate per minute (HR) systolic blood pressure (SAP) diastolic blood pressure (DAP) peripheral oxygen saturation (SpO2) and simultaneous block and contralateral Perfusion index: PI, Plethysmographic index of variability: PVI values were recorded by measuring baseline, post-block 1st, 5th, 10th, 15th, and 20th values. After the measurements, the patients with successful block were presented to surgery. Patients without complications after surgery were transferred to the service.

ELIGIBILITY:
Inclusion Criteria:

* ASA classification (American Society of Anesthesiologists) I-II score
* no contraindications for block
* patient's acceptance

Exclusion Criteria:

* Pediatric patients
* pregnant patients
* patients with peripheral arterial disease
* renal failure
* liver failure
* coagulation disorder

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: patients who will undergo upper-term surgery
Sampling Method: Probability Sample
Enrollment: 2 (Actual)
Dates: Start 2021-01-01 (Actual); Primary Completion 2021-03-01 (Actual); Study Completion 2021-05-01 (Actual)

PRIMARY OUTCOMES:
Perfusion index: PI | 10 WEEK
  monitoring, both upper extremities Perfusion index: PI, (The probe of a MasimoRadical 7, MasimoCorp. Irvine, CA, USA) were performed.

SECONDARY OUTCOMES:
Plethysmographic variability index: PVI | 10 WEEK
  monitoring, both upper extremities , Plethysmographic variability index: PVI, (The probe of a MasimoRadical 7, MasimoCorp. Irvine, CA, USA) were performed.

OTHER OUTCOMES:
hemoglobin HGB, | 10 WEEK
  monitoring, both upper extremities hemoglobin HGB, (The probe of a MasimoRadical 7, MasimoCorp. Irvine, CA, USA) were performed.

CONTACTS AND LOCATIONS:
Locations (1):
- Malatya Eğitim Ve Araştirma Hastanesi, Malatya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No